CLINICAL TRIAL: NCT07339072
Title: Temporal Interference Methods for Non-invasive Deep Brain Stimulation
Brief Title: Temporal Interference Methods for Non-invasive Deep Brain Stimulation, Study 1.2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Brown, PHD, Professor of Pyschological and Brain Science, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 26941, Study 1.2; 1R21MH140210-01 (NIH)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: Temporal Interference; fMRI; BOLD Signal; Cognitive Control; Dorsal Anterior Cingulate Cortex; Non-invasive deep brain stimulation; Neurostimulation

STUDY DESIGN:
Intervention Model Description: This study uses a within-subject crossover design. Participants receive both active temporal interference (TI) stimulation and sham stimulation, in both "on" and "off" conditions during fMRI scanning. The order of active vs. sham stimulation and the order of on vs off conditions is counterbalanced across participants. Beat frequency, electrode placement, and behavioral paradigm vary by sub-study (e.g., reward-related tasks targeting the nucleus accumbens, cognitive control and decision-making tasks targeting the dorsal anterior cingulate cortex). For Study 1.2, two temporal interference beat frequencies (5 Hz and 10 Hz) will be evaluated for their effects on the nucleus accumbens.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- NAcc 5 Hz TI Active, then NAcc 5 Hz TI Sham, then NAcc 10 Hz TI Active, then NAcc 10 Hz TI Sham (Active Comparator): Participants in this arm receive temporal interference (TI) electrical stimulation targeting the nucleus accumbens using two pairs of carbon fiber electrodes in the following order: 5 Hz TI Active, 5 Hz TI Sham, 10 Hz TI Active, then 10 Hz TI Sham.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Sham
- NAcc 5 Hz TI Sham, then NAcc 5 Hz TI Active, then NAcc 10 Hz TI Sham, then NAcc 10 Hz TI Active (Active Comparator): Participants in this arm receive temporal interference (TI) electrical stimulation targeting the nucleus accumbens using two pairs of carbon fiber electrodes in the following order: 5 Hz TI Sham, 5 Hz TI Active, 10 Hz TI Sham, then 10 Hz TI Active.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Sham
- NAcc 10 Hz TI Sham, then NAcc 10 Hz TI Active, then NAcc 5 Hz TI Sham, then NAcc 5 Hz TI Active (Active Comparator): Participants in this arm receive temporal interference (TI) electrical stimulation targeting the nucleus accumbens using two pairs of carbon fiber electrodes in the following order: 10 Hz TI Sham, 10 Hz TI Active, 5 Hz TI Sham, then 5 Hz TI Active.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Sham
- NAcc 10 Hz TI Active, then NAcc 10 Hz TI Sham, then NAcc 5 Hz TI Active, then NAcc 5 Hz TI Sham (Active Comparator): Participants in this arm receive temporal interference (TI) electrical stimulation targeting the nucleus accumbens using two pairs of carbon fiber electrodes in the following order: 10 Hz TI Active, 10 Hz TI Sham, 5 Hz TI Active, then 5 Hz TI Sham.
  Interventions: Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Sham; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Active; Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Sham

INTERVENTIONS:
Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Active — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using alternating current frequencies at up to 2 mA per electrode. For the NAcc 5 Hz TI Active condition, one channel will deliver 2000 Hz and the other 2005 Hz, producing a 5 Hz beat frequency that focally stimulates deep brain regions without activating overlying cortex. Stimulation is administered in 2-minute on / 2-minute off cycles with a 30-second ramp up and ramp down beginning at the start of each 2-minute period.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc 5 Hz TI Sham — Same setup as the 5 Hz TI Active condition, except that the stimulation immediately ramps down as soon as it reaches 2 mA after ramp up, producing a sham condition.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Active — Non-invasive electrical brain stimulation delivered through two sets of scalp electrodes using alternating current frequencies at up to 2 mA per electrode. For the NAcc 10 Hz TI Active condition, one channel will deliver 2000 Hz and the other 2010 Hz, producing a 10 Hz beat frequency that focally stimulates deep brain regions without activating overlying cortex. Stimulation is administered in 2-minute on / 2-minute off cycles with a 30-second ramp up and ramp down beginning at the start of each 2-minute period.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation
Device: Temporal Interference (TI) Electrical Stimulation - NAcc 10 Hz TI Sham — Same setup as the 10 Hz TI Active condition, except that the stimulation immediately ramps down as soon as it reaches 2 mA after ramp up, producing a sham condition.
  Other Names: TI Electrical Neurostimulation; TI Neurostimulation

SUMMARY:
In its totality, this grant aims to develop a line of research using temporal interference (TI) electrical neurostimulation technology to understand the causal role of deep brain structures in cognition. In the short term, the investigators aim to validate and characterize the effects of TI on brain activity as measured by fMRI and demonstrate its ability to focally stimulate deep brain regions without affecting overlying cortex. In the longer term, investigators aim to use these data to resolve longstanding debates about the function of deeper brain regions and lay the foundation for future clinical applications of TI for treating addiction, Obsessive-Compulsive Disorder (OCD), Parkinson's disease, and other disorders involving deep brain dysfunction. The grant supports 2 distinct aims, each of which will be evaluated through a series of independent studies.

DETAILED DESCRIPTION:
Through the grant's duration, the investigators hypothesize that temporal interference (TI) electrical neurostimulation will be well tolerated and effective at focally manipulating deep brain activity as measured by functional MRI (fMRI) BOLD signals. The investigators will investigate whether TI stimulation can increase BOLD activity in targeted deep brain regions including the nucleus accumbens (NAcc) and dorsal anterior cingulate cortex (dACC), and whether this stimulation can influence cognitive functions controlled by these regions. TI works by applying alternating currents of slightly different frequencies through multiple electrode pairs, creating an interference pattern that can stimulate deep brain regions without significantly affecting superficial cortical areas. This method is similar to traditional transcranial direct current stimulation (tDCS), however TI can stimulate deeper brain structures that tDCS cannot reach effectively. The study is broken up into two main aims with multiple sub-studies. In Aim 1, the investigators will characterize the effects of TI on fMRI BOLD signals, test different beat frequencies, and compare TI effects in the nucleus accumbens versus dorsal anterior cingulate cortex. In Aim 2, the investigators will apply TI to the dorsal anterior cingulate cortex to test causal theories about its role in cognitive control, conflict monitoring, risk avoidance, and foraging behavior using established cognitive tasks while subjects undergo fMRI scanning.

Study 1.2 (Aim 1, Study 12) will test the ability to focally activate the nucleus accumbens without activating the overlying cortex, and also its effects on functional connectivity. Healthy subjects (n=30) will present for a single study visit during which they will be placed in the fMRI scanner and administered a temporal interference protocol. Specifically, subjects will have four pairs of carbon fiber electrodes attached to the scalp with conductive gel. They will receive one 8-minute block of stimulation at 2mA per electrode pair. The stimulation sequence will be 2 minutes on, 2 minutes off, 2 minutes on, and 2 minutes off with 30 second ramp up and ramp down beginning at the start of each 2-minute period. For Study 1.2, two TI beat frequencies will be evaluated: 5 Hz (produced by channels at 2000 Hz and 2005 Hz) and 10 Hz (produced by channels at 2000 Hz and 2010 Hz). Each beat frequency will have an Active block (30-second ramp to 2 mA, 2 min on / 2 min off cycles) and a matching Sham block where the stimulation immediately ramps down as soon as it reaches 2 mA after ramp up. The order of blocks and whether the "on" or "off" condition occurs first will be counterbalanced across subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50
* Must have at least a 6th grade education
* Ability to speak and read English for all phases

Exclusion Criteria:

* Currently taking psychotropic medications for ADHD, other mental illness, or medications for cancer
* History of epilepsy or seizure disorders
* History of migraines or other neurological syndromes
* History of AIDS (due to potential cognitive deficits)
* History of head trauma or cognitive impairments
* Personal experiences consistent with symptoms of psychosis (e.g., hallucinations, delusions of control or special powers)
* History of skull defects (e.g., holes bored into the skull or known cranial fissures)
* Metal implants in the head or under the scalp
* Does not meet fMRI safety screening criteria (e.g., metal implants in the body, permanent jewelry, tattoos on the head or neck)
* Uses an intrauterine device (IUD) for birth control and cannot provide documentation to verify MRI safety
* Pregnancy (self-reported; no pregnancy test administered)
* Weight over 440 lbs (scanner weight limit)
* Presence of pacemakers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-03 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
Change in brain activity in the nucleus accumbens during 5 Hz versus 10 Hz temporal interference stimulation | During fMRI scan on study day (approximately 60 minutes)
  Brain activity in the nucleus accumbens will be measured using functional magnetic resonance imaging (fMRI) during temporal interference (TI) stimulation at 5 Hz compared to 10 Hz. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal, which reflects changes in neural activity. Higher BOLD values indicate stronger brain activation.

SECONDARY OUTCOMES:
Change in brain activity in the nucleus accumbens during active versus sham stimulation at 5 Hz | During fMRI scan on study day (approximately 60 minutes)
  Brain activity in the nucleus accumbens will be measured using fMRI during active versus sham temporal interference stimulation at a 5 Hz beat frequency. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal.
Change in brain activity in the nucleus accumbens during active versus sham stimulation at 10 Hz | During fMRI scan on study day (approximately 60 minutes)
  Brain activity in the nucleus accumbens will be measured using fMRI during active versus sham temporal interference stimulation at a 10 Hz beat frequency. Activity will be reported as the percent change in blood-oxygen-level-dependent (BOLD) signal.
Change in brain connectivity between the nucleus accumbens and other brain regions during temporal interference stimulation | During fMRI scan on study day (approximately 60 minutes)
  Functional connectivity between the nucleus accumbens and other brain regions will be measured using fMRI-based analyses during active versus sham temporal interference stimulation. Higher correlation values indicate stronger communication between brain regions. The primary test statistic will be the whole-brain psycho-physiological interaction (PPI) between nucleus accumbens BOLD activity and stimulation condition.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua W Brown, PhD, Principal Investigator — Indiana University, Bloomington
Locations (1):
- Indiana University Bloomington, Imaging Research Facility, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Violante IR, Alania K, Cassara AM, Neufeld E, Acerbo E, Carron R, Williamson A, Kurtin DL, Rhodes E, Hampshire A, Kuster N, Boyden ES, Pascual-Leone A, Grossman N. Non-invasive temporal interference electrical stimulation of the human hippocampus. Nat Neurosci. 2023 Nov;26(11):1994-2004. doi: 10.1038/s41593-023-01456-8. Epub 2023 Oct 19. Erratum In: Nat Neurosci. 2023 Dec;26(12):2252. doi: 10.1038/s41593-023-01517-y. PMID 37857775
- [Background] Modak P, Fine J, Colon B, Need E, Cheng H, Hulvershorn L, Finn P, Brown JW. Temporal interference electrical neurostimulation at 20 Hz beat frequency leads to increased fMRI BOLD activation in orbitofrontal cortex in humans. Brain Stimul. 2024 Jul-Aug;17(4):867-875. doi: 10.1016/j.brs.2024.07.014. Epub 2024 Jul 24. PMID 39059712
- [Background] Grossman N, Bono D, Dedic N, Kodandaramaiah SB, Rudenko A, Suk HJ, Cassara AM, Neufeld E, Kuster N, Tsai LH, Pascual-Leone A, Boyden ES. Noninvasive Deep Brain Stimulation via Temporally Interfering Electric Fields. Cell. 2017 Jun 1;169(6):1029-1041.e16. doi: 10.1016/j.cell.2017.05.024. PMID 28575667
- See also: Lab website for study. The Cognitive Control Lab aims to understand the neural mechanisms of goal-directed behavior, using a combination of fMRI, computational neural modeling, and neurostimulation methods in healthy and clinical human populations. — https://ccsrv1.psych.indiana.edu/cclab/
- See also: Project details for the NIMH-funded study on temporal interference stimulation, including abstract, funding, and key personnel. — https://reporter.nih.gov/project-details/11119339